CLINICAL TRIAL: NCT00338689
Title: Childhood Obesity - Programming by Infant Nutrition
Brief Title: European Childhood Obesity Project: Early Programming by Infant Nutrition?
Acronym: CHOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Prof. Dr. Dr., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00389
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Infant Development
Keywords: infant formula; protein content; growth; obesity; breast feeding
MeSH Terms: conditions — Obesity; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower protein formula (Experimental): Intervention: Infant formula with relatively low protein content (1.25 g/ 100 ml) during the first year of life; described as "Lower protein formula"
  Interventions: Dietary Supplement: Lower protein formula; Higher protein formula
- Higher protein formula (Placebo Comparator): Intervention: Infant formula with a relatively high protein content (2.05 g/ 100 ml) during the first year of life; described as "Higher protein formula"
  Interventions: Dietary Supplement: Lower protein formula; Higher protein formula
- Breastfed reference group (No Intervention): Non-randomized breastfed group of infants at least 3 months exclusively breastfed

INTERVENTIONS:
Dietary Supplement: Lower protein formula; Higher protein formula — During the intervention phase of the study, which is from inclusion in the study (latest age 2 weeks) until age 12 months, two experimental infant formulae with different protein content are fed to the enrolled infants; Lower protein formula and Higher protein formula. Additional a breastfed observational group without any intervention is included.
  Arms: Higher protein formula; Lower protein formula

SUMMARY:
Primary hypothesis to be tested:

Early protein intake predicts infant growth and later risk of childhood obesity.

* Childhood obesity is a major public health problem and is an identified priority concern for the health care. Infants fed formula are more likely to become obese than breastfed infants. The higher protein content of infant formulae, compared with breast milk, could be a causal factor.
* The study will in a multicentre intervention trial on newborn infants investigate whether feeding infant formulae, which differ in their level of milk proteins, can influence the risk of later childhood obesity. The trial will take place in five countries with different habitual total protein intakes to increase the range of protein intakes
* The investigators will study body composition, hormonal status, protein metabolism and anthropometric markers of childhood obesity. The whole cohort will be followed up until age 18 years, to assess the long term impact on the prevalence of obesity.
* The investigators will explore the impact of consumer (parental) attitudes to, and perceptions of, different practices of infant feeding in relation to infant behaviour (satisfaction, crying, sleep duration). This consumer science information will help improve the understanding of consumer (infants and parents) acceptance of and preference for foods that contribute to healthy diets.
* If a relationship between early dietary protein intake and later childhood obesity risk is confirmed, it offers possibilities for the prevention of obesity, for improving advice given to parents and for developing nutritionally improved dietary products for infants.

DETAILED DESCRIPTION:
Obesity has become a global epidemic and is a major health challenge for children and ado-lescents in industrialised countries, with a high and steadily increasing prevalence. Individual obesity risk is strongly influenced by genetic disposition and lifestyle factors. But in addition, there are clear indications that metabolic events during pre- and postnatal development mark-edly modulate obesity risk in later life, known as metabolic programming. Epidemiological studies and animal experiments suggest a causal relationship between nutrition early in life and the risk of later obesity, e.g. breast feeding seems to reduce the risk of obesity.

One factor clearly different between breast and formula fed infants is the protein intake, and thus in the Childhood Obesity Project the influence of this factor will be tested by feeding in double blind random-ised clinical trial two formulas with different protein content (7.3 % vs. 12 % of energy) to infants from five European countries (Belgium, Germany, Italy, Poland, Spain). Protein supply via formula is defined for the first year of life, while additional food is only recorded. Until the age of 2 years the growth and development of the infants is followed by frequent stand-ardised measurements and data on socio-economic status, parental attitudes and medical his-tory are collected. The available data will be evaluated in respect to the influence of protein intake and all the other factors on anthropometric markers for later obesity. This seems justi-fied as the weight and length growth until the age of 2 years have been shown to predict the body mass index with 14 years, suggesting that this is a suitable and very early indicator for overweight later in life.

Furthermore, differences between the participating countries will be studied with the aim to identify further environmental factors influencing obesity risk. On a long term base it is planned to follow the study participants via mailed questionnaires until the age of eight years to validate the risk estimators in a huge well defined population.

Primary objectives:

* To test the influence of the protein content of the infant formula fed during the first year of life on growth until the age of two years (main outcome measures: length and weight velocity).
* First year protein intake predicts later risk of childhood obesity ('Early protein hypothe-sis'). Primary outcome measure: BMI at the age of 8 years.
* Protein intake in the first year of life is associated to long-term metabolic outcomes: BMI and Body Composition at 18 years

Secondary objectives:

* Evaluation of the effects of different habitual protein intakes with traditional complemen-tary feeding regimes in infants in 5 European countries.
* Examination of the relationship between different types of infant feeding regimes with respect to Beikost on an early anthropometric markers of later obesity development.
* Investigation of effects of these infant feeding regimes on body composition, energy ex-penditure, protein metabolism, renal function and size, leptin and its binding protein and on IGF-1.
* Exploration of consumer attitudes and infant feeding practices in relation to parental obe-sity status.
* Investigation of the mediation of the relationship between diet and later growth via bio-chemical parameters, which might become detectable by the plasma concentrations of the corresponding compounds at the age of 6 months.
* Investigation of the effects of infant behaviour (esp. crying, sleeping and feeding behav-iour) on development of obesity.
* Comparison of the weight and length development to a non randomised cohort of breast-fed infants.
* Measurement of the effects of dietary regimes on body composition measured by stable dilution techniques (subgroup only).
* Measurement of the effects of dietary regimes on total energy expenditure and exploration of relationships between TEE, body composition and obesity risk (subgroup only).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks
* Appropriate for gestational age (above 10th percentile,Lubchenko)
* Age of the mother at least 18 years
* Singleton pregnancies
* Residence in the study area
* Maternal command of the language

Exclusion Criteria:

* Gestational diabetes
* Major malformations (of the child) which might interfere with nutrition or growth
* Hormonal or metabolic diseases of the mother or the child, drug addiction during pregnancy

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1678 (Actual)
Dates: Start 2002-10; Primary Completion 2006-08 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Body mass index BMI: derived from measured body height (m) and body weight (kg) as body weight / height² | At age 11 years and 18 years
  Body height (cm) will be determined with calibrated clinical equipment Body weight (kg) will be determined with calibrated clinical equipment BMI calculated

SECONDARY OUTCOMES:
Dietary intake | At 1-9,12,18 and 24 months, at 3, 4, 5, 6, 8, 11, 18 years
  3 day dietary protocols and food frequency questionnaires, (at 11and 18 years only EFPQ)
Blood parameters | At age 6 months, 5.5 years, 8 years, 11 and 18 years
  Partially: Plasma amino acids, hormones, NEFAs, Polar-Lipids, triglycerides
Physical activity | At age 2, 4, 6, 8, 11 years (questionnaires), at 6, 8, 11, 18 years accelerometer
  Physical activity questionnaire and sensewear accelerometer data
Body composition | at 3, 6, 12, 24 months, biannually from 3 to 6 years, at 7,8,11, 18 years
  Skinfold measurements at all time points, additionally bioelectrical impedance at 5, 5.5, 6, 7,8 11 and years, partly additionaly air displacement plethysmography at 18 years
Urine markers | At 6 months, 5.5, 8, 11 and 18 years
  Uric acid, urea, creatinine, calcium secretion, C-peptide (not at 18 years)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Ludwig-Maximilians-Universitaet
Locations (5):
- CHC St. Vincent, Liège / Universite Libre de Bruxelles, Liège, Belgium
- Ludwig-Maximilians-Universitaet, München, Germany
- Universita degli Studi di Milano, Milan, Italy
- Children´s Memorial Healzj Institute, Warsaw, Poland
- Universitat Rovira i Virgili, Tarragona, Spain

REFERENCES:
- [Derived] Totzauer M, Escribano J, Closa-Monasterolo R, Luque V, Verduci E, ReDionigi A, Langhendries JP, Martin F, Xhonneux A, Gruszfeld D, Socha P, Grote V, Koletzko B; European Childhood Obesity Trial Study Group. Different protein intake in the first year and its effects on adiposity rebound and obesity throughout childhood: 11 years follow-up of a randomized controlled trial. Pediatr Obes. 2022 Dec;17(12):e12961. doi: 10.1111/ijpo.12961. Epub 2022 Jul 25. PMID 36355369
- [Derived] Jaeger V, Koletzko B, Luque V, Ferre N, Gruszfeld D, Gradowska K, Verduci E, Zuccotti GV, Xhonneux A, Poncelet P, Grote V. Distribution of energy and macronutrient intakes across eating occasions in European children from 3 to 8 years of age: The EU Childhood Obesity Project Study. Eur J Nutr. 2023 Feb;62(1):165-174. doi: 10.1007/s00394-022-02944-6. Epub 2022 Aug 5. PMID 35930067
- [Derived] Xhonneux A, Langhendries JP, Martin F, Seidel L, Albert A, Dain E, Totzauer M, Grote V, Luque V, Closa-Monasterolo R, Dionigi AR, Verduci E, Gruszfeld D, Socha P, Koletzko B; European Childhood Obesity Trial Study group. Parental Perception of Body Weight Status of Their 8-year-old Children: Findings from the European CHOP Study. Matern Child Health J. 2022 Jun;26(6):1274-1282. doi: 10.1007/s10995-021-03334-w. Epub 2022 Jan 1. PMID 34982337
- [Derived] Guerlich K, Gruszfeld D, Czech-Kowalska J, Ferre N, Closa-Monasterolo R, Martin F, Poncelet P, Verduci E, Koletzko B, Grote V. Sleep duration and problem behaviour in 8-year-old children in the Childhood Obesity Project. Eur Child Adolesc Psychiatry. 2022 Mar;31(3):519-527. doi: 10.1007/s00787-021-01731-8. Epub 2021 Feb 24. PMID 33624130
- [Derived] Aumueller N, Gruszfeld D, Gradowska K, Escribano J, Ferre N, Martin F, Poncelet P, Verduci E, ReDionigi A, Koletzko B, Grote V. Influence of total sugar intake on metabolic blood markers at 8 years of age in the Childhood Obesity Project. Eur J Nutr. 2021 Feb;60(1):435-442. doi: 10.1007/s00394-020-02229-w. Epub 2020 May 6. PMID 32377804
- [Derived] Aumueller N, Gruszfeld D, Gradowska K, Escribano J, Ferre N, Rousseaux D, Hoyos J, Verduci E, ReDionigi A, Koletzko B, Grote V. Associations of sugar intake with anthropometrics in children from ages 2 until 8 years in the EU Childhood Obesity Project. Eur J Nutr. 2020 Sep;59(6):2593-2601. doi: 10.1007/s00394-019-02107-0. Epub 2019 Oct 23. PMID 31642983
- [Derived] Schwarzfischer P, Gruszfeld D, Socha P, Luque V, Closa-Monasterolo R, Rousseaux D, Moretti M, Mariani B, Verduci E, Koletzko B, Grote V. Longitudinal analysis of physical activity, sedentary behaviour and anthropometric measures from ages 6 to 11 years. Int J Behav Nutr Phys Act. 2018 Dec 7;15(1):126. doi: 10.1186/s12966-018-0756-3. PMID 30526600
- [Derived] Schwarzfischer P, Gruszfeld D, Stolarczyk A, Ferre N, Escribano J, Rousseaux D, Moretti M, Mariani B, Verduci E, Koletzko B, Grote V. Physical Activity and Sedentary Behavior From 6 to 11 Years. Pediatrics. 2019 Jan;143(1):e20180994. doi: 10.1542/peds.2018-0994. Epub 2018 Dec 3. PMID 30509928
- [Derived] Totzauer M, Luque V, Escribano J, Closa-Monasterolo R, Verduci E, ReDionigi A, Hoyos J, Langhendries JP, Gruszfeld D, Socha P, Koletzko B, Grote V; European Childhood Obesity Trial Study Group. Effect of Lower Versus Higher Protein Content in Infant Formula Through the First Year on Body Composition from 1 to 6 Years: Follow-Up of a Randomized Clinical Trial. Obesity (Silver Spring). 2018 Jul;26(7):1203-1210. doi: 10.1002/oby.22203. PMID 29932518
- [Derived] Gomes D, Luque V, Xhonneux A, Verduci E, Socha P, Koletzko B, Berger U, Grote V. A simple method for identification of misreporting of energy intake from infancy to school age: Results from a longitudinal study. Clin Nutr. 2018 Jun;37(3):1053-1060. doi: 10.1016/j.clnu.2017.05.003. Epub 2017 Jun 1. PMID 28780991
- [Derived] Schwarzfischer P, Weber M, Gruszfeld D, Socha P, Luque V, Escribano J, Xhonneux A, Verduci E, Mariani B, Koletzko B, Grote V. BMI and recommended levels of physical activity in school children. BMC Public Health. 2017 Jun 24;17(1):595. doi: 10.1186/s12889-017-4492-4. PMID 28645324
- [Derived] Closa-Monasterolo R, Zaragoza-Jordana M, Ferre N, Luque V, Grote V, Koletzko B, Verduci E, Vecchi F, Escribano J; Childhood Obesity Project Group. Adequate calcium intake during long periods improves bone mineral density in healthy children. Data from the Childhood Obesity Project. Clin Nutr. 2018 Jun;37(3):890-896. doi: 10.1016/j.clnu.2017.03.011. Epub 2017 Mar 16. PMID 28351509
- [Derived] Zaragoza-Jordana M, Closa-Monasterolo R, Luque V, Ferre N, Grote V, Koletzko B, Pawellek I, Verduci E, ReDionigi A, Socha J, Stolarczyk A, Poncelet P, Rousseaux D, Escribano J; Childhood Obesity Project Group. Micronutrient intake adequacy in children from birth to 8 years. Data from the Childhood Obesity Project. Clin Nutr. 2018 Apr;37(2):630-637. doi: 10.1016/j.clnu.2017.02.003. Epub 2017 Feb 9. PMID 28238467
- [Derived] Kirchberg FF, Harder U, Weber M, Grote V, Demmelmair H, Peissner W, Rzehak P, Xhonneux A, Carlier C, Ferre N, Escribano J, Verduci E, Socha P, Gruszfeld D, Koletzko B, Hellmuth C; European Childhood Obesity Trial Study Group. Dietary protein intake affects amino acid and acylcarnitine metabolism in infants aged 6 months. J Clin Endocrinol Metab. 2015 Jan;100(1):149-58. doi: 10.1210/jc.2014-3157. PMID 25368978
- [Derived] Weber M, Grote V, Closa-Monasterolo R, Escribano J, Langhendries JP, Dain E, Giovannini M, Verduci E, Gruszfeld D, Socha P, Koletzko B; European Childhood Obesity Trial Study Group. Lower protein content in infant formula reduces BMI and obesity risk at school age: follow-up of a randomized trial. Am J Clin Nutr. 2014 May;99(5):1041-51. doi: 10.3945/ajcn.113.064071. Epub 2014 Mar 12. PMID 24622805
- [Derived] Rzehak P, Grote V, Lattka E, Weber M, Gruszfeld D, Socha P, Closa-Monasterolo R, Escribano J, Giovannini M, Verduci E, Goyens P, Martin F, Langhendries JP, Demmelmair H, Klopp N, Illig T, Koletzko B; European Childhood Obesity Trial Study Group. Associations of IGF-1 gene variants and milk protein intake with IGF-I concentrations in infants at age 6 months - results from a randomized clinical trial. Growth Horm IGF Res. 2013 Oct;23(5):149-58. doi: 10.1016/j.ghir.2013.05.002. Epub 2013 Jun 22. PMID 23800627
- [Derived] Luque V, Escribano J, Grote V, Ferre N, Koletzko B, Gruszfeld D, Socha P, Langhendries JP, Goyens P, Closa-Monasterolo R; European Childhood Obesity Project. Does insulin-like growth factor-1 mediate protein-induced kidney growth in infants? A secondary analysis from a randomized controlled trial. Pediatr Res. 2013 Aug;74(2):223-9. doi: 10.1038/pr.2013.87. Epub 2013 May 24. PMID 23708690
- [Derived] Luque V, Escribano J, Mendez-Riera G, Schiess S, Koletzko B, Verduci E, Stolarczyk A, Martin F, Closa-Monasterolo R. Methodological approaches for dietary intake assessment in formula-fed infants. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):320-7. doi: 10.1097/MPG.0b013e3182779a60. PMID 23443063
- [Derived] Closa-Monasterolo R, Ferre N, Luque V, Zaragoza-Jordana M, Grote V, Weber M, Koletzko B, Socha P, Gruszfeld D, Janas R, Xhonneux A, Dain E, Scaglioni S, Escribano J; Childhood Obesity Project Study Group. Sex differences in the endocrine system in response to protein intake early in life. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1920S-1927S. doi: 10.3945/ajcn.110.001123. Epub 2011 Nov 16. PMID 22089446
- [Derived] Grote V, Schiess SA, Closa-Monasterolo R, Escribano J, Giovannini M, Scaglioni S, Stolarczyk A, Gruszfeld D, Hoyos J, Poncelet P, Xhonneux A, Langhendries JP, Koletzko B; European Childhood Obesity Trial Study Group. The introduction of solid food and growth in the first 2 y of life in formula-fed children: analysis of data from a European cohort study. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1785S-1793S. doi: 10.3945/ajcn.110.000810. Epub 2011 Sep 14. PMID 21918213
- [Derived] Socha P, Grote V, Gruszfeld D, Janas R, Demmelmair H, Closa-Monasterolo R, Subias JE, Scaglioni S, Verduci E, Dain E, Langhendries JP, Perrin E, Koletzko B; European Childhood Obesity Trial Study Group. Milk protein intake, the metabolic-endocrine response, and growth in infancy: data from a randomized clinical trial. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1776S-1784S. doi: 10.3945/ajcn.110.000596. Epub 2011 Aug 17. PMID 21849603
- [Derived] Koletzko B, von Kries R, Closa R, Escribano J, Scaglioni S, Giovannini M, Beyer J, Demmelmair H, Gruszfeld D, Dobrzanska A, Sengier A, Langhendries JP, Rolland Cachera MF, Grote V; European Childhood Obesity Trial Study Group. Lower protein in infant formula is associated with lower weight up to age 2 y: a randomized clinical trial. Am J Clin Nutr. 2009 Jun;89(6):1836-45. doi: 10.3945/ajcn.2008.27091. Epub 2009 Apr 22. PMID 19386747